CLINICAL TRIAL: NCT05705869
Title: Targeted Assessment in High-Risk paTients With dIAbetes to ideNtify Undiagnosed Heart Failure (TARTAN-HF)
Brief Title: Targeted Assessment in High-Risk paTients With dIAbetes to ideNtify Undiagnosed Heart Failure
Acronym: TARTAN-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GN22CA228
Record Dates: First submitted 2022-12-21; First posted 2023-01-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Diabetes Mellitus; Type 1 Diabetes; Type 2 Diabetes; Cardiovascular Diseases
Keywords: Screening; Primary Care; Secondary Care; NT-proBNP; Echocardiogram; Diagnostic Pathway
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine care arm (No Intervention): Patients in this arm will undergo routine diabetes care. They will be managed and followed up as per routine clinical care. They will be remotely monitored for heart failure events electronically. Quality of life questionnaires (Kansas City Cardiomyopathy Questionnaire-12 and EQ-5D) will be collected.
- Investigational arm (Experimental): Patients in this arm will have a blood sample taken to measure N-terminal prohormone of B-type natriuretic peptide (NT-proBNP).
  In addition to this, routine blood samples, an ECG, body measurements, patient reported outcomes and observations will be recorded.
  Further blood and urine samples will be collected and stored within Glasgow University storage facilities for future measurement of relevant biomarkers and for use in future ethically approved research.
  Patients with an elevated NT-proBNP (≥125 pg/mL) will undergo a full cart-based transthoracic echocardiogram along with a clinical examination for signs of HF and a HF symptom assessment. Patients will then also undergo a handheld echocardiogram with a CE-marked handheld point of care EchoNous Kosmos echocardiogram device.
  Patients who are classified as having heart failure (HFrEF, HFmrEF, or HFpEF) will be managed according to the latest version of European Society of Cardiology guidelines.
  Interventions: Diagnostic Test: NT-proBNP

INTERVENTIONS:
Diagnostic Test: NT-proBNP — NT-proBNP will be measured in all participants in the Investigational arm. If the level of the NT-proBNP is elevated (≥125pg/mL) participants will undergo a full cart-based transthoracic echocardiogram along with a clinical examination for signs of HF and a HF symptom assessment. Participants with HF identified will be referred to their local HF clinic for ongoing management.
  Arms: Investigational arm

SUMMARY:
This is a prospective, multicentre, unblinded, randomised, controlled trial. The primary aim is to assess a targeted screening strategy to detect undiagnosed heart failure in high-risk patients with diabetes.

DETAILED DESCRIPTION:
This is a prospective, multicentre, unblinded, randomised, controlled trial. The primary aim is to assess a targeted screening strategy to detect undiagnosed heart failure in high-risk patients with diabetes.

Participants will be recruited from the diabetes service in two NHS health boards in Scotland; NHS Greater Glasgow and Clyde and NHS Lanarkshire. At the point of recruitment and consent, patients will be randomised to one of two arms:

1. "Routine care arm" - patients in this arm will undergo routine diabetes care. They will be managed and followed up as per routine clinical care. They will be remotely monitored for HF events electronically. Quality of life questionnaires (Kansas City Cardiomyopathy Questionnaire-12 and EQ-5D) will be completed electronically through CASTOR program in this arm (with the option of paper versions for participants who can not use CASTOR).

   OR
2. "Investigational arm" - patients in this arm will have a blood sample taken to measure N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) using a Roche assay. In addition to this, blood samples for haemoglobin, creatinine, HbA1c, cholesterol profile, liver function tests and eGFR will be collected. Quality of life questionnaires (Kansas City Cardiomyopathy Questionnaire-12 and EQ-5D) will be completed electronically through CASTOR program in this arm (with the option of paper versions for participants who can not use CASTOR).

All patients in this arm will also have an ECG and basic body measurements and observations measured. Further venous blood samples will be collected and stored within Glasgow University storage facilities for future measurement of relevant biomarkers and for use in future ethically approved research. Urine samples will also be collected for measurement of urine albumin:creatinine ratio and for future measurement of relevant biomarkers and use in future ethically approved research.

Patients with an elevated Roche NT-proBNP (≥125 pg/mL) will undergo a full cart-based transthoracic echocardiogram along with a clinical examination for signs of HF and a HF symptom assessment. A British Society of Echocardiography minimum dataset will be obtained, and report created.

Patients will then also undergo a handheld echocardiogram with a UKCE-marked handheld point of care (POC) EchoNous Kosmos echocardiogram device. The handheld echocardiogram images will be acquired by a British Society of Echocardiography accredited operator. The US2.ai algorithm (which is also UKCE marked) will generate an AI-automated echocardiogram report.

Patients who are classified as having heart failure (HFrEF, HFmrEF, or HFpEF) will be managed according to the latest version of European Society of Cardiology guidelines for the diagnosis and treatment of acute and chronic heart failure. The results of the cart-based echocardiogram will be used during the determination of the presence or absence of HF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥40 years of age
* Informed consent
* An established diagnosis of diabetes (type 1 or type 2)
* At least one additional risk factor for heart failure:

  1. Coronary artery disease (either a previous documented type 1 myocardial infarction or coronary artery bypass grafting or percutaneous coronary intervention or documented stenosis of an epicardial coronary artery [>50% left main or >70% left anterior descending, circumflex or right coronary artery])
  2. Persistent or permanent atrial fibrillation (not paroxysmal atrial fibrillation)
  3. Previous ischemic or embolic stroke
  4. Peripheral arterial disease (previous surgical or percutaneous revascularisation or a documented stenosis greater than 50% of a major peripheral arterial vessel).
  5. Chronic kidney disease (defined as an estimated glomerular filtration rate <60mL/min/1.73m2 or eGFR 60-90mL/min/1.73m2 and UACR >300mg/g).
  6. Regular loop diuretic use (any dose at any dosing interval) for >30 days.
  7. COPD (evidenced by one of the following; PFTs showing airway obstruction, diagnosis by respiratory physician, CT scan reporting presence of emphysema or treatment with national guideline-advocated COPD therapy).

Exclusion Criteria:

* Inability to give informed consent e.g., due to significant cognitive impairment.
* Previous documented diagnosis of heart failure.
* Echocardiogram or NT-proBNP interpreted as excluding heart failure within 12 months.
* Currently receiving scheduled renal replacement therapy.
* Anyone who, in the investigators' opinion, is not suitable to participate in the trial for other reasons e.g., a diagnosis which may compromise survival over the study period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of heart failure within 6 months | 6 months

SECONDARY OUTCOMES:
Diagnosis of HFrEF within 6 months | 6 months
People diagnosed with HFrEF receiving GDMT within 6 months | 6 months

OTHER OUTCOMES:
Diagnosis of HFmrEF within 6 months | 6 months
Diagnosis of HFpEF within 6 months | 6 months
People diagnosed with HFmrEF and HFpEF receiving SGLT2i therapy within 6 months | 6 months
Diagnosis of asymptomatic left ventricular dysfunction (LVEF≤40%) within 6 months | 6 months
Time to first heart failure hospitalisation at 1 year | 1 year
Time to first heart failure hospitalisation at 2 years | 2 years
Time to first heart failure hospitalisation at 5 years | 5 years
All-cause mortality at 1 year | 1 year
All-cause mortality at 2 years | 2 years
All-cause mortality at 5 years | 5 years
Time to first occurence of any components of the following clinical composite 1) heart failure hospitalisation 2) all-cause mortality at 1 year | 1 year
Time to first occurence of any components of the following clinical composite 1) heart failure hospitalisation 2) all-cause mortality at 2 years | 2 years
Time to first occurence of any components of the following clinical composite 1) heart failure hospitalisation 2) all-cause mortality at 5 years | 5 years
The incremental cost-effectiveness ratio (ICER) will be expressed as incremental costs/life-year gained | 5 years
he accuracy of handheld echocardiography with AI-automated reporting compared to full cart-based echocardiogram and manual reporting for the measurement of LVEF (%) | 6 months
The number of patients in the NT-proBNP/echocardiography group with echocardiographic features of potential amyloid as assessed by the US2.ai algorithm report conclusion of "amyloid to be considered" | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Petrie, MbChB, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Queen Elizabeth University Hospital, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No